CLINICAL TRIAL: NCT04418154
Title: Neoadjuvant Anthracycline Followed by Toripalimab Combined With Nab-paclitaxel in Patients With Early Triple-negative Breast Cancer
Brief Title: Neoadjuvant Dose-dense EC Followed by ABX With PD-1 for Triple Negative Breast Cancer Patients
Acronym: NeoTENNIS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiong Wu, Professor, Department of Breast Surgery Vice President, Cancer Hospital, Fudan University, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N027
Record Dates: First submitted 2020-05-25; First posted 2020-06-05 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: Programmed Death-1
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Albumin-Bound Paclitaxel; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EC-ABX/PD-1 (Experimental): Patients who are treated with epirubicin hydrochloride andcyclophosphamide followed by nanoparticlealbumin-bound paclitaxel and Toripalimab
  Interventions: Drug: epirubicin hydrochloride; Drug: Cyclophosphamide; Drug: Albumin bound paclitaxel; Drug: Toripalimab

INTERVENTIONS:
Drug: epirubicin hydrochloride — Take epirubicin hydrochloride (90mg/m2, d1) every 14 days as one cycle for 4 cycles with cyclophosphamide, followed by nanoparticlealbumin-bound paclitaxel and Toripalimab.
Drug: Cyclophosphamide — Take cyclophosphamide (600mg/m2, d1) every 14 days as one cycle for 4 cycles with epirubicin hydrochloride, followed by nanoparticlealbumin-bound paclitaxel and Toripalimab.
Drug: Albumin bound paclitaxel — Take nanoparticlealbumin-bound paclitaxel (125mg/m2, d1) per week for 3 weeks as one cycle for 4 cycles with Toripalimab, following epirubicin hydrochloride and cyclophosphamide.
Drug: Toripalimab — Take Toripalimab (240mg, d1) every 3 weeks as one cycle for 4 cycles with nanoparticlealbumin-bound paclitaxel, following epirubicin hydrochloride and cyclophosphamide.

SUMMARY:
This study is to evaluate the efficacy and safety for dose-dense epirubicin hydrochloride with cyclophosphamide followed by nanoparticlealbumin-bound paclitaxel with PD-1 in neoadjuvant therapy for patients with triple-negative breast cancer, and to explore the predictive value of biological markers for the treatment.

DETAILED DESCRIPTION:
This study is an open single arm study, which would undergo optimal two stage designs. 60 patients who are diagnosed with triple-negative breast cancer would have dose-dense epirubicin hydrochloride with cyclophosphamide followed by nanoparticlealbumin-bound paclitaxel with PD-1 regimen for neoadjuvant therapy if they meet the eligibility criteria. The regimen is as follows: epirubicin hydrochloride (90mg/m2, d1) plus cyclophosphamide (600mg/m2, d1) every 14 days as one cycle for 4 cycles, followed by nanoparticlealbumin-bound paclitaxel (125mg/m2, d1) per week for 3 weeks as one cycle for 4 cycles, and Toripalimab (240mg, d1) every 3 weeks as one cycle for 4 cycles. pathological complete response would be the primary endpoint. The change of biological markers and safety of the regimen would also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old, female.
* Patients with histologically confirmed unilateral primary invasive breast cancer who meet the criteria of cT2-4NanyM0.
* Patients with ER negative and PR negative by immunohistochemistry (IHC), and HER-2 negative disease. HER2-negative disease was defined as follows: disease whose HER-2 is 1+ or negative by IHC, or fluorescence in situ hybridization (FISH) is negative if IHC is 2+.
* According to the RECIST 1.1 criteria, there is at least one measurable objective lesion.
* Eastern Cooperative Oncology Group (ECOG) performance score 0-1.
* Baseline left ventricular ejection fraction (LVEF) is greater than or equal to (>/=) 55%.
* Bone marrow function is required as follows: neutrophils are more than or equal to (>/=) 1.5×109/L, platelets more than or equal to (>/=) 100×109/L, and hemoglobin more than or equal to (>/=) 90g/L.
* Hepatic and renal function are required as follows: serum creatinine is less than or equal to (</=) 1.5 times of upper limits of normal (ULN), aspartate transaminase (AST) and alanine aminotransferase (ALT) less than or equal to (</=) 2.5 times of ULN, and total bilirubin less than or equal to (</=) 1.5 times of ULN or </= 2.5 times of ULN if patient is with Gilbert's syndrome.
* With good compliance with the planned treatment, are able to understand the follow-up procedures of this study and sigh the informed consent form.

Signed informed consent.

Exclusion Criteria:

* Received radiotherapy, chemotherapy, surgery or other targeted and immunotherapy for triple-negative breast cancer before enrollment.
* With heart disease classified as New York Heart Association class (NYHA) grade II or above (including grade II) are identified by the investigator.
* With severe systemic infection or those with other serious illnesses.
* Known to be allergic or intolerant to chemotherapy drugs or their excipients.
* With a history of autoimmune diseases or those using glucocorticoids or immunosuppressive drugs.
* With known active stage of HBV or HCV infection or hepatitis B DNA ≥500, or patients with chronic abnormal liver function.
* With a history of abnormal thyroid function.
* With grade ≥ 2 peripheral neuropathy.
* With a clear history of neurological or mental disorders, including epilepsy or dement.
* Previous non-breast malignancy within 5 years prior to study entry excluding healed cervical carcinoma in situ and non-melanoma skin cancer.
* History of other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ and non-melanoma skin cancer.
* Pregnancy or lactation, and patients of childbearing potential who refuse to use adequate contraception during the course of this study.
* Prior participation in other studies within 30 days prior to the administration of the first dose of the investigational drug.
* Patients who are deemed to be unsuitable for this study by investigators.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Pathologic complete response (tpCR) | Immediately after the surgery
  Defined as no residual invasive cancer cells are found in the pathological examination of breast and axillary lymph node; if only residual in situ cancer cells are present in the surgical specimens, it can also be considered as achieving a pathological complete response.

SECONDARY OUTCOMES:
Breast pathologic complete response (bpCR: ypT0/is) rate | Immediately after the surgery
  Defined as the absence of invasive cancer cells in breast.
Objective response rate (ORR) | Immediately after the surgery
  Defined as the proportion of patients with a complete or partial response by MRI.
Breast conservative surgery rate | Immediately after the surgery
  Defined as the percentage of patients who undergo breast-conserving surgery after neoadjuvant therapy, out of the total number of evaluable cases.
Event-free survival (EFS) | Approximately 3 years
  Defined as the time from the date of the first study dose to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Adverse events (AEs) | During this period between the start of randomization and the last visit, approximately 3 years
  Refer to any untoward medical occurrence in a study subject administered an investigational product which does not necessarily have a causal relationship with the treatment. AE is assessed according to the NCI-CTCAE 5.0.
Change in immune-related tissue biomarkers | At baseline, at the end of first 2 cycles (each cycle is 14 days) and immediately after the surgery
  The proportion of Tumor-infiltrating lymphocytes (TILs) is evaluated through HE staining. Immunohistochemical staining of PD-1, PD-L1, AR, CD8, and FOXC1) is performed. TILs, PD1, PD-L1, AR, CD8, and FOXC1 in tumor samples by biopsy at baseline, at the end of Cycle 2 and by surgery immediately after surgery would be evaluated by HE or immune staining.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] He M, Hao S, Ma L, Xiu B, Yang B, Wang Z, Xue J, Chi Y, Xiong M, Chen J, Huang X, Liu X, Wu S, Xiao Q, Huang Y, Shui R, Cao A, Li J, Di G, Yang W, Hu X, Liu G, Yu K, Jiang Y, Wang Z, Shao Z, Wu J. Neoadjuvant anthracycline followed by toripalimab combined with nab-paclitaxel in patients with early triple-negative breast cancer (NeoTENNIS): a single-arm, phase II study. EClinicalMedicine. 2024 Jun 28;74:102700. doi: 10.1016/j.eclinm.2024.102700. eCollection 2024 Aug. PMID 39045544